CLINICAL TRIAL: NCT02148341
Title: Implementation of the Hospital to Home (H2H) Heart Failure Initiative
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Paul Heidenreich, Staff Physician, VA Palo Alto Health Care System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SDP-09-160
Record Dates: First submitted 2013-02-12; First posted 2014-05-28 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2013-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Community of Practice Facilitation (Experimental): Medical Centers assigned to this arm will recieive the communtiy of practice facilitation. In this process we will contact existing members of the community of practice (called the Heart Failure Network) at the facility as well as attempt to identify new providers and other staff at the facility with an interest in improving heart failure care. The facilitation includes: describing the national H2H program, providing talking points and strategies for local providers to obtain support from their local facility to initiate local projects related to H2H, providing a forum for successful sites to describe how they initiated projects to sites yet to initiate projects.
  Interventions: Other: Community of Practice Facilitation
- Usual Care (Experimental): Medical centers in this arm will hear of H2H through usual routs (calls with facilty Directors and Chiefs of staff).
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Community of Practice Facilitation
  Arms: Community of Practice Facilitation
Other: Usual Care
  Arms: Usual Care

SUMMARY:
This study determines if a community of practice of clinicians and quality improvement specialists can be used to implement a national quality initiative known as Hospital to Home (H2H). This quality initative is designed to reduced readmission rates for patients with heart failure or heart attack by improving the transition of care upon discharge.

ELIGIBILITY:
Inclusion Criteria:

* VA medical centers are the unit of randomization. A medical center will be included if had at least 20 patients discharged with a principal diagnosis of heart failure in 2008

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2010-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
H2H enrollment | 6 months
  H2H enrollment by the facility as determined by the H2H program of the American College of Cardiology and Institute for Healthcare Improvement

SECONDARY OUTCOMES:
quality improvement programs initiated due to H2H | 6 months
  A new quality improvement initiated that addressess one of the 3 areas of H2H focus. These include, medication reconcilliation, early follow-up after discharge, and symptom recognition.

CONTACTS AND LOCATIONS:
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States